CLINICAL TRIAL: NCT05899556
Title: A Comprehensive View of Patient Experiences of Individuals Participating in Pulmonary Fibrosis Clinical Study
Brief Title: Pinpointing the Factors Affecting Clinical Study Experiences of Pulmonary Fibrosis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83217345
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in clinical trials usually favors a particular demographic group. But there is limited research available to explain what research attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of pulmonary fibrosis patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future pulmonary fibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of pulmonary fibrosis
* Ability to understand the study procedures, benefits and risks, and sign a written informed consent document.

Exclusion Criteria:

* Enrolled in another research study
* Inability to provide written informed consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary fibrosis who are actively participating in a clinical research, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of pulmonary fibrosis patients who decide to participate in a clinical study | 3 months
Rate of patients who remain in an pulmonary fibrosis clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aiello M, Bertorelli G, Bocchino M, Chetta A, Fiore-Donati A, Fois A, Marinari S, Oggionni T, Polla B, Rosi E, Stanziola A, Varone F, Sanduzzi A. The earlier, the better: Impact of early diagnosis on clinical outcome in idiopathic pulmonary fibrosis. Pulm Pharmacol Ther. 2017 Jun;44:7-15. doi: 10.1016/j.pupt.2017.02.005. Epub 2017 Feb 28. PMID 28257817
- [Background] Glass DS, Grossfeld D, Renna HA, Agarwala P, Spiegler P, DeLeon J, Reiss AB. Idiopathic pulmonary fibrosis: Current and future treatment. Clin Respir J. 2022 Feb;16(2):84-96. doi: 10.1111/crj.13466. Epub 2022 Jan 10. PMID 35001525
- [Background] O'Riordan TG, Smith V, Raghu G. Development of novel agents for idiopathic pulmonary fibrosis: progress in target selection and clinical trial design. Chest. 2015 Oct;148(4):1083-1092. doi: 10.1378/chest.14-3218. PMID 26020856

DOCUMENTS (1):
  • Informed Consent Form (2023-06-02): https://cdn.clinicaltrials.gov/large-docs/56/NCT05899556/ICF_000.pdf